CLINICAL TRIAL: NCT01952327
Title: Investigation Into the Automated Drainage of Recurrent Effusions From the Pleural Space in Thoracic Malignancy.
Acronym: ADEPT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sequana Medical N.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-AAR-008
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- plueurapump (Other): Implantation of pleurapump system
  Interventions: Device: The pleurapump system

INTERVENTIONS:
Device: The pleurapump system — Implantation of the pleurapump system

SUMMARY:
This is a research study examining the safety of a new, automated pump for the drainage of fluid in the chest cavity which is caused by cancer (also known as malignant pleural effusion, or MPE). The purpose of the trial is to assess whether the new pleurapump device is safe and effective in the management of patients with MPE. The study will try to identify what kind of problems may arise from using the device, how often they happen, and how severe they are if they occur.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Recurrent pleural effusion due malignancy Malignant pleural effusions are defined as either Fluid in the context of histocytologically confirmed pleural malignancy, or pleural fluid in the context of histocytologically confirmed malignancy elsewhere, with no other clear cause for the effusion.
3. 1 or more therapeutic procedures for pleural fluid drainage prior to enrolment.
4. Written informed consent
5. Ability to comply with study procedures and ability to operate the device
6. Expected survival of more than 3 months after device insertion

Exclusion Criteria:

1. Haemothorax
2. Purulent pleural effusion
3. Significant pleural fluid septation or loculation on thoracic ultrasound or cross-sectional imaging
4. Obstructive uropathy or any bladder anomaly which might contraindicate implantation of the device.
5. Pregnant females or females anticipating pregnancy during study period.
6. Patients currently enrolled in another interventional clinical study
7. Concurrently implanted with any other Active Implantable Medical Device, including, but not limited to cardiac pacemaker or cardioverter defibrillator.
8. Major comorbidity which, in the opinion of the principal investigator, is likely to significantly decrease life expectancy, increase anaesthetic risk, or lead to device removal (e.g. moderate to severe congestive heart failure, significant valvular heart disease, persistent immunosuppression, etc.)
9. Other contraindication to general anaesthesia
10. Other contraindication to procedure (e.g. uncorrectable bleeding diathesis, infection or malignant involvement over proposed insertion site)
11. Significant renal impairment, as determined by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of device, procedure and therapy related serious adverse events. | 3 months
  Incidence and severity of device, procedure and therapy related serious adverse events.

SECONDARY OUTCOMES:
Efficacy of treatment as assessed by the volume of fluid removed | 3 months
  Efficacy of treatment as assessed by the volume of fluid removed by the pump
Need for further intervention to manage pleural fluid (on the side of the intervention) | 3 months
  Need for further intervention to manage pleural fluid (on the side of the intervention), including therapeutic thoracentesis of greater than 100mls, insertion of an indwelling catheter, insertion of an intercostal drain for fluid management, or thoracoscopy.
Subjective thoracic pain on the side of the intervention | 3 months
  Subjective thoracic pain on the side of the intervention (measured using VAS score)
Subjective abdominal pain | 3 months
  Subjective abdominal pain (measured using VAS score)
Subjective breathlessness | 3 months
  Subjective breathlessness (measured using VAS score)
Quality of life | 3 months
  Quality of life, measured using EQ-5D health questionnaires
Costs of health resource use | 3 months
  Costs of health resource use over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Nick Maskell, MD, Principal Investigator — Dept. of Respiratory Medicine, Southmead Hospital, Bristol, BS10 5NB, United Kingdom
Locations (2):
- Oncologie Thoracique - Maladies de la Plèvre - Pneumologie Interventionnelle, Hôpital Nord, Marseille, France
- Dept. of Respiratory Medicine, Southmead Hospital, Bristol, United Kingdom